CLINICAL TRIAL: NCT06411769
Title: Evidence-based Intervention to Improve Walking Engagement in El Paso, Texas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: U01MD019289 (NIH); 7U01MD019289-02 (NIH)
Record Dates: First submitted 2024-04-26; First posted 2024-05-13 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Activity Trackers; Physical Activity
Keywords: Walking Challenge; Moderate-to-Vigorous-Physical Activity; Evidence-based; Employer-based
MeSH Terms: conditions — Motor Activity | interventions — Schools

STUDY DESIGN:
Intervention Model Description: This study will draw upon Sequential, Multiple Assignment, Randomized Trials (SMART) design to reduce barriers for both individuals and worksites to improve responsiveness to individual performance. The investigators are using the Consolidated Framework for Implementation Research (CFIR) across all project activities to establish proof-of-concept and improve the quality of behavioral intervention delivery to disparate populations on the U.S.-Mexico border and other similar regions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase 1. 50K4LIfe Only (Experimental): Walking Challenge only
  Interventions: Behavioral: 50K4LIfe
- Phase 1. 50K4Life + SMS Text Messages (Experimental): Walking Challenge + SMS Messages
  Interventions: Behavioral: 50K4LIfe; Behavioral: SMS Text Messaging
- Phase 2. 50K4LIfe + Individual (Experimental): Walking Challenge + Individual level interventions.
  Interventions: Behavioral: 50K4LIfe; Behavioral: Individual
- Phase 2. 50K4LIfe + School (Experimental): Walking Challenge + School-level interventions
  Interventions: Behavioral: 50K4LIfe; Behavioral: School
- Phase 2. 50K4Life + SMS Text Messages + Individual (Experimental): Walking Challenge + SMS Messages + Individual level interventions
  Interventions: Behavioral: 50K4LIfe; Behavioral: SMS Text Messaging; Behavioral: Individual
- Phase 2. 50K4Life + SMS Text Messages + Schools (Experimental): Walking Challenge + SMS Messages + School-level interventions
  Interventions: Behavioral: 50K4LIfe; Behavioral: SMS Text Messaging; Behavioral: School
- Phase 2. Walking Challenge only (Experimental): Participants meeting the step goal in Phase 1(WC only) will continue into Phase 2 without change.
  Interventions: Behavioral: 50K4LIfe
- Phase 2. Walking Challenge + SMS Text Messages (Experimental): Participants meeting their step goal in Phase 1 (WC + SMS Text Messages) will continue into Phase 2 without change.
  Interventions: Behavioral: 50K4LIfe; Behavioral: SMS Text Messaging

INTERVENTIONS:
Behavioral: 50K4LIfe — This intervention will consist of the Walking Challenge only.
Behavioral: SMS Text Messaging — In this intervention, participants will received notifications onto the Pathverse app
  Arms: Phase 1. 50K4Life + SMS Text Messages; Phase 2. 50K4Life + SMS Text Messages + Individual; Phase 2. 50K4Life + SMS Text Messages + Schools; Phase 2. Walking Challenge + SMS Text Messages
Behavioral: Individual — In this Phase 2 individual-level intervention, participants will receive remote education modules and one-to-one monthly phone-based coaching.
  Arms: Phase 2. 50K4LIfe + Individual; Phase 2. 50K4Life + SMS Text Messages + Individual
Behavioral: School — In this Phase 2 school-level intervention, participants will receive group educational sessions, school environmental modifications (floor distance markings, signage in corridors and breakrooms, promotional items), and participate in work time/weekend group walks/hikes.
  Arms: Phase 2. 50K4LIfe + School; Phase 2. 50K4Life + SMS Text Messages + Schools

SUMMARY:
The investigators will test if the 50,000 for Life (50K4Life) is effective at improving walking engagement in school employees in 30 public schools by delivering a two-phased adaptive intervention to improve walking engagement in school workers in 30 public schools. In Phase 1, all study schools will be randomly assigned to a 50K4Life only, or 50K4Life + SMS Text Messaging group.

In Phase 2, non-responder schools will be randomly assigned to one of two 6-month adaptive treatments: a) an individual-level intervention that includes remote education modules (REM) and one-to-one monthly phone-based coaching, or, b) a school-level intervention that includes group educational sessions, school environmental modifications (floor distance markings, signage in corridors and breakrooms, promotional items), and work time/weekend group walks/hikes. The schools that 50% or more participants who achieve 50,000 steps in one week will continue with the Phase 1 condition. Intervention strategies will be coordinated by health educators and managed using the Pathverse app. Data collection will occur at baseline, 8 weeks (Phase 2 randomization decision point), 8 months (immediate post intervention), 12 months (4 months post-intervention), and 18 months (10 months post-intervention) for a total of 18 months of study participation.

DETAILED DESCRIPTION:
Mexican Americans who live in the U.S.-Mexico border region suffer disproportionately from preventable cardiometabolic diseases. Regular brisk walking is an effective measure in regulating metabolic processes and preventing disease. Employer-based wellness programs are promising strategies to address this public health problem because of the opportunity to take advantage of workplace environments to improve opportunities for walking engagement while also addressing barriers associated with inactivity. Employer-based walking programs have not been widely tested on the U.S.-Mexico border. A clustered Sequential Multiple Assignment Randomized Trial (SMART) will be conducted to determine the effectiveness of an employer-based walking challenge intervention- 50,000 for Life (50K4Life)- in improving brisk walking engagement (at least 7,000 steps/day) among school district employees. The proposed intervention strategies are based on the walking interventions conducted by the Principal Investigator(s) in El Paso and behavioral, environmental and worksite interventions by the Co-Investigators. The trial will include 30 randomly selected public schools with predominantly Mexican American employees from El Paso County area school districts. The intervention strategies in 50K4Life will be in two phases: 1) 50K4Life vs. 50K4Life + SMS text messaging and 2) Individual vs. School level adaptation for campuses with a low response to the initial intervention phase. The investigators hypothesize that walking challenges with multilevel capacity building and adaptations based on intervention response will lead to improved adherence to PA guidelines. This proposed socioecological model-based study leverages resources through Hispanic Serving Institutions (HSI) from Texas and expertise in employer-based workplace interventions from the University of Georgia (UGA) based on the partner's accumulative work to address the disparity in PA and advance health equity in the Mexican American population. As part of the intervention evaluation, the PIs will conduct a process evaluation and cost-effectiveness to provide insight into cost and scalability. This study will provide needed information on optimizing the implementation of evidence-based behavioral interventions to improve walking engagement among Mexican Americans living in the U.S.-Mexico border region.

ELIGIBILITY:
Inclusion Criteria:

* A school is eligible if it is located within one of the four target school districts
* adult 18 years or older
* full-time school-based school district employee
* not pregnant and able to walk without physical limitations or assistive device
* willing to wear our Fitbit tracking device or use their own tracking device for 18 months
* own a smartphone
* willingness to use a personal smartphone for tracking activity related to the Fitbit tracker, access online intervention content, and receive text messages.

Exclusion Criteria:

* Works at more than one school
* Does not work on a district school campus
* schools that previously participated in walking challenges

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Daily Step Count | Daily, Weekly up to 18 months.
  The Pathverse app synced with an activity tracker will be used to collect daily step counts. The goal is for teams (schools) to have 50% of their staff with an average weekly steps > 50,000.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness (CVF) | Baseline, 8 weeks, 8 months, 12, months 18 months up to 18 months.
  The heart rate/minute at the end of the YMCA 3-minute submaximal bench-stepping test will be used to assess the level of CVF associated with increased PA.
Weight | Baseline, 8 weeks, 8 months, 12 months, 18 months up to 18 months.
  Weight (to the nearest 0.1 kg) will be collected using a portable scale
Height | Baseline
  Height (measured to the nearest 0.1 cm) will be obtained using a stadiometer.
Body Mass Index | Baseline, 8 weeks, 8 months, 12 months, 18 months up to 18 months.
  Body Mass Index (BMI) will be calculated as weight (kg)/height squared (m2).
Waist Circumference | Baseline, 8 weeks, 8 months, 12 months, 18 months up to 18 months.
  Waist circumference will be measured at the midway between the iliac crests and the lower ribs.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Salinas, Ph.D., LMSW, Principal Investigator — University of Texas, El Paso
Locations (1):
- University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hourdou ML, Besson F, Michel G. Studies on the biosynthesis of beta-amino acids, the lipid moiety of iturins A, in Bacillus subtilis. J Antibiot (Tokyo). 1988 Feb;41(2):207-11. doi: 10.7164/antibiotics.41.207. PMID 3128514
- [Background] Tucker JM, Welk GJ, Beyler NK. Physical activity in U.S.: adults compliance with the Physical Activity Guidelines for Americans. Am J Prev Med. 2011 Apr;40(4):454-61. doi: 10.1016/j.amepre.2010.12.016. PMID 21406280
- [Background] Karstoft K, Clark MA, Jakobsen I, Muller IA, Pedersen BK, Solomon TP, Ried-Larsen M. The effects of 2 weeks of interval vs continuous walking training on glycaemic control and whole-body oxidative stress in individuals with type 2 diabetes: a controlled, randomised, crossover trial. Diabetologia. 2017 Mar;60(3):508-517. doi: 10.1007/s00125-016-4170-6. Epub 2016 Dec 9. PMID 27942800
- [Background] Bailey MM, Coller RK, Pollack Porter KM. A qualitative study of facilitators and barriers to implementing worksite policies that support physical activity. BMC Public Health. 2018 Sep 27;18(1):1145. doi: 10.1186/s12889-018-6045-x. PMID 30261871
- [Background] Garne-Dalgaard A, Mann S, Bredahl TVG, Stochkendahl MJ. Implementation strategies, and barriers and facilitators for implementation of physical activity at work: a scoping review. Chiropr Man Therap. 2019 Oct 9;27:48. doi: 10.1186/s12998-019-0268-5. eCollection 2019. PMID 31624537
- [Background] Sedani A, Stover D, Coyle B, Wani RJ. Assessing Workplace Health and Safety Strategies, Trends, and Barriers through a Statewide Worksite Survey. Int J Environ Res Public Health. 2019 Jul 11;16(14):2475. doi: 10.3390/ijerph16142475. PMID 31336749
- [Background] Wu S, Fisher-Hoch SP, Reninger B, McCormick JB. Meeting or Exceeding Physical Activity Guidelines is Associated with Reduced Risk for Cancer in Mexican-Americans. Am J Cancer Prev. 2016;4(1):1-7. doi: 10.12691/ajcp-4-1-1. Epub 2016 Jan 29. PMID 28529961
- [Background] Salinas JJ, Valenzuela R, Sheen J, Carlyle M, Gay J, Morales A. An ORBIT Phase 1: Design study of a citywide employer-based walking challenges in a predominantly Mexican American metropolitan area. J Health Psychol. 2022 Mar;27(4):961-973. doi: 10.1177/1359105320977650. Epub 2020 Dec 20. PMID 33345634
- [Background] Saadiq S, Valenzuela R, Wang J, Yin Z, Parra-Medina D, Gay J, Salinas JJ. Walking Engagement in Mexican Americans Who Participated in a Community-Wide Step Challenge in El Paso, TX. Int J Environ Res Public Health. 2021 Dec 2;18(23):12738. doi: 10.3390/ijerph182312738. PMID 34886463
- [Background] Salinas JJ, McDaniel M, Parra-Medina D. The Role of Social Support and the Neighborhood Environment on Physical Activity in Low-income, Mexican-American Women in South Texas. J Prev Med Public Health. 2018 Sep;51(5):234-241. doi: 10.3961/jpmph.18.052. Epub 2018 Jul 25. PMID 30286595
- [Background] Parra-Medina D, Hilfinger Messias DK. Promotion of Physical Activity Among Mexican-Origin Women in Texas and South Carolina: An Examination of Social, Cultural, Economic, and Environmental Factors. Quest. 2011 Feb;63(1):100-117. doi: 10.1080/00336297.2011.10483668. PMID 21731409
- [Background] Mitchell MS, Orstad SL, Biswas A, Oh PI, Jay M, Pakosh MT, Faulkner G. Financial incentives for physical activity in adults: systematic review and meta-analysis. Br J Sports Med. 2020 Nov;54(21):1259-1268. doi: 10.1136/bjsports-2019-100633. Epub 2019 May 15. PMID 31092399
- [Background] Marteau TM, Ashcroft RE, Oliver A. Using financial incentives to achieve healthy behaviour. BMJ. 2009 Apr 9;338:b1415. doi: 10.1136/bmj.b1415. No abstract available. PMID 19359291
- [Background] Weinstock J, Petry NM. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults. Ann Intern Med. 2016 Oct 18;165(8):599. doi: 10.7326/L16-0281. No abstract available. PMID 27750317
- [Background] Meng L, Wolff MB, Mattick KA, DeJoy DM, Wilson MG, Smith ML. Strategies for Worksite Health Interventions to Employees with Elevated Risk of Chronic Diseases. Saf Health Work. 2017 Jun;8(2):117-129. doi: 10.1016/j.shaw.2016.11.004. Epub 2016 Dec 2. PMID 28593067
- [Background] Mehta S, Dimsdale J, Nagle B, Holub CK, Woods C, Barquera S, Elder JP. Worksite interventions: improving lifestyle habits among Latin American adults. Am J Prev Med. 2013 May;44(5):538-42. doi: 10.1016/j.amepre.2013.01.015. PMID 23597820
- [Background] Chandrasekaran B, Rao CR, Davis F, Arumugam A. SMART STEP - SMARTphone-driven exercise and pedometer-based STEP intervention to promote physical activity among desk-based employees: Study protocol for a three-arm cluster randomized controlled trial. Work. 2021;69(4):1229-1245. doi: 10.3233/WOR-213544. PMID 34366306
- [Background] Freak-Poli R, Cumpston M, Albarqouni L, Clemes SA, Peeters A. Workplace pedometer interventions for increasing physical activity. Cochrane Database Syst Rev. 2020 Jul 21;7(7):CD009209. doi: 10.1002/14651858.CD009209.pub3. PMID 32700325
- [Background] Wolfenden L, Goldman S, Stacey FG, Grady A, Kingsland M, Williams CM, Wiggers J, Milat A, Rissel C, Bauman A, Farrell MM, Legare F, Ben Charif A, Zomahoun HTV, Hodder RK, Jones J, Booth D, Parmenter B, Regan T, Yoong SL. Strategies to improve the implementation of workplace-based policies or practices targeting tobacco, alcohol, diet, physical activity and obesity. Cochrane Database Syst Rev. 2018 Nov 14;11(11):CD012439. doi: 10.1002/14651858.CD012439.pub2. PMID 30480770
- [Background] Stephenson A, McDonough SM, Murphy MH, Nugent CD, Mair JL. Using computer, mobile and wearable technology enhanced interventions to reduce sedentary behaviour: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2017 Aug 11;14(1):105. doi: 10.1186/s12966-017-0561-4. PMID 28800736
- [Background] Jung J, Cho I. Promoting Physical Activity and Weight Loss With mHealth Interventions Among Workers: Systematic Review and Meta-analysis of Randomized Controlled Trials. JMIR Mhealth Uhealth. 2022 Jan 21;10(1):e30682. doi: 10.2196/30682. PMID 35060913
- [Background] Muir SD, Silva SSM, Woldegiorgis MA, Rider H, Meyer D, Jayawardana MW. Predictors of Success of Workplace Physical Activity Interventions: A Systematic Review. J Phys Act Health. 2019 Aug 1;16(8):647-656. doi: 10.1123/jpah.2018-0077. PMID 31203701
- [Background] Salinas JJ, Parra-Medina D. Physical activity change after a promotora-led intervention in low-income Mexican American women residing in South Texas. BMC Public Health. 2019 Jun 20;19(1):782. doi: 10.1186/s12889-019-7105-6. PMID 31221117
- [Background] Yin Z, Errisuriz VL, Evans M, Inupakutika D, Kaghyan S, Li S, Esparza L, Akopian D, Parra-Medina D. A Digital Health Intervention for Weight Management for Latino Families Living in Rural Communities: Perspectives and Lessons Learned During Development. JMIR Form Res. 2020 Aug 20;4(8):e20679. doi: 10.2196/20679. PMID 32726748
- [Background] Yin Z, Lesser J, Paiva KA, Zapata J Jr, Moreno-Vasquez A, Grigsby TJ, Ryan-Pettes SR, Parra-Medina D, Estrada V, Li S, Wang J. Using Mobile Health Tools to Engage Rural Underserved Individuals in a Diabetes Education Program in South Texas: Feasibility Study. JMIR Mhealth Uhealth. 2020 Mar 24;8(3):e16683. doi: 10.2196/16683. PMID 32207694
- [Background] Parra-Medina D, Mojica C, Liang Y, Ouyang Y, Ramos AI, Gomez I. Promoting Weight Maintenance among Overweight and Obese Hispanic Children in a Rural Practice. Child Obes. 2015 Aug;11(4):355-63. doi: 10.1089/chi.2014.0120. Epub 2015 May 7. PMID 25950140
- [Background] Gay JL, Buchner DM. Ethnic disparities in objectively measured physical activity may be due to occupational activity. Prev Med. 2014 Jun;63:58-62. doi: 10.1016/j.ypmed.2014.02.015. Epub 2014 Feb 28. PMID 24589439
- [Background] Gay JL, Buchner DM, Smith J. Occupational Physical Activity Opposes Obesity: A Cross-Sectional Modern Replication of the Morris 1953 London Busmen Study. J Occup Environ Med. 2019 Mar;61(3):177-182. doi: 10.1097/JOM.0000000000001489. PMID 30395010
- [Background] Gay JL, Buchner DM, Smith J, He C. An examination of compensation effects in accelerometer-measured occupational and non-occupational physical activity. Prev Med Rep. 2017 Aug 5;8:55-59. doi: 10.1016/j.pmedr.2017.07.013. eCollection 2017 Dec. PMID 28879071
- [Background] Gay JL, Saunders RP, Rees-Punia E, Dowda M, van den Berg AE. Role of Organizational Support on Implementation of an Environmental Change Intervention to Improve Child Fruit and Vegetable Intake: a Randomized Cross-Over Design. Prev Sci. 2019 Nov;20(8):1211-1218. doi: 10.1007/s11121-019-01043-z. PMID 31468247
- [Background] Wang J, Sereika SM, Chasens ER, Ewing LJ, Matthews JT, Burke LE. Effect of adherence to self-monitoring of diet and physical activity on weight loss in a technology-supported behavioral intervention. Patient Prefer Adherence. 2012;6:221-6. doi: 10.2147/PPA.S28889. Epub 2012 Mar 22. PMID 22536058
- [Background] Wang J, Chu CF, Li C, Hayes L, Siminerio L. Diabetes Educators' Insights Regarding Connecting Mobile Phone- and Wearable Tracker-Collected Self-Monitoring Information to a Nationally-Used Electronic Health Record System for Diabetes Education: Descriptive Qualitative Study. JMIR Mhealth Uhealth. 2018 Jul 26;6(7):e10206. doi: 10.2196/10206. PMID 30049667
- [Background] Valenzuela R, Morales A, Sheen J, Rangel S, Salinas JJ. The Implementation of Evidence-Based Obesity Education Curricula to Prevent Cancer in a Predominantly Mexican-American Community on the U.S.-Mexico Border. J Cancer Educ. 2023 Feb;38(1):215-224. doi: 10.1007/s13187-021-02101-3. Epub 2021 Oct 8. PMID 34623603
- [Background] Wang J, Cai C, Padhye N, Orlander P, Zare M. A Behavioral Lifestyle Intervention Enhanced With Multiple-Behavior Self-Monitoring Using Mobile and Connected Tools for Underserved Individuals With Type 2 Diabetes and Comorbid Overweight or Obesity: Pilot Comparative Effectiveness Trial. JMIR Mhealth Uhealth. 2018 Apr 10;6(4):e92. doi: 10.2196/mhealth.4478. PMID 29636320
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Ramirez M, Wu S, Beale E. Designing a Text Messaging Intervention to Improve Physical Activity Behavior Among Low-Income Latino Patients With Diabetes: A Discrete-Choice Experiment, Los Angeles, 2014-2015. Prev Chronic Dis. 2016 Dec 22;13:E171. doi: 10.5888/pcd13.160035. PMID 28005532
- [Background] Morton K, Sutton S, Hardeman W, Troughton J, Yates T, Griffin S, Davies M, Khunti K, Eborall H. A Text-Messaging and Pedometer Program to Promote Physical Activity in People at High Risk of Type 2 Diabetes: The Development of the PROPELS Follow-On Support Program. JMIR Mhealth Uhealth. 2015 Dec 15;3(4):e105. doi: 10.2196/mhealth.5026. PMID 26678750